CLINICAL TRIAL: NCT03550027
Title: Indwelling Pleural Catheter for Trapped Lung: a Pilot Study for Power Calculation of a Randomized Controlled Trial Comparing Pleurocath® Versus PleurX®)
Brief Title: Indwelling Pleural Catheter for Trapped Lung
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R 574/17 - IEO 607
Record Dates: First submitted 2018-03-21; First posted 2018-06-08 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2018-06

CONDITIONS: Pleura; Effusion
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PleurX (Experimental): Positioning of Pleurx drainage during surgical exploration if lung does not reinflate
  Interventions: Device: PleurX
- Pleurocath (Experimental): Positioning of Pleur o cath drainage during surgical exploration if lung does not reinflate
  Interventions: Device: Pleurocath

INTERVENTIONS:
Device: PleurX — Positioning of drainage PleurX
  Arms: PleurX
Device: Pleurocath — Positioning of drainage Pleurocath
  Arms: Pleurocath

SUMMARY:
Malignant pleural effusion (MPE) is a complication of almost any site of primary cancer as well as primary tumors of the pleura. Half of MPE patients have non-expendable trapped lungs not suitable for talc pleurodesis. Indwelling pleural catheters (IPCs), however, can be used in this cohort of patients, bringing about an improvement in dyspnea and quality of life (QOL).

The aim of this study is to obtain pilot data - comparing patients receiving two different types of indwelling pleural catethers normally used in clinical practice (10 patients receiving Pleurocath® and 10 patients receiving PleurX®) - for power calculation of a Randomized Controlled Trial comparing two different drainages for MPE trapped lung.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, with a clinical confident diagnosis of symptomatic malignant pleural effusion, enrolled for VATS exploration but not amenable of VATS talc poudrage because of trapped lung (patients with only partial expansion however receiving talc poudrage, but needing permanent pleural cathetes, are also eligible)

Exclusion Criteria:

* - Age younger than 18 years
* Expected survival of less than 3 months
* Chylothorax
* Total white blood cell count less than 1000/microL
* Pregnancy or lactating mothers
* Irreversible bleeding diathesis
* Irreversible visual impairment
* Contraindications to general anesthesia
* Poor general clinical conditions ( ECOG PS >=2)
* Patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) range 0 (no pain) - 100 (maximum pain) | Post operative day 4th
  Thoracic pain
Visual Analog Scale (VAS) range 0 (no dyspnea) - 100 (maximim dyspnea) | Post operative day 4th
  Dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Petrella, MD, PhD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided